CLINICAL TRIAL: NCT00085488
Title: En Vivo Matured Dendritic Cell Therapy in Patients With Melanoma
Brief Title: Vaccine Therapy in Treating Patients With Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000370802; DMS-9935; DMS-14862
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2005-10

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage III melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — FANG vaccine

INTERVENTIONS:
Biological: autologous tumor cell vaccine
Biological: therapeutic autologous dendritic cells

SUMMARY:
RATIONALE: Vaccines made from a patient's dendritic cells and tumor cells may make the body build an immune response to kill tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vaccine therapy in treating patients with stage III or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the dose-limiting toxicity and the maximum tolerated dose of autologous dendritic cells pulsed with autologous tumor cell lysate in patients with stage III or IV melanoma.
* Determine the safety and tolerability of this therapy in these patients.

Secondary

* Determine the immune response, in terms of the type and degree of T-cell proliferation and delayed-type hypersensitivity responses, in patients treated with this therapy.

OUTLINE: This is a dose-escalation, pilot study.

Patients undergo leukapheresis for the collection of peripheral blood mononuclear cells (PBMC) on days -9, 19, and 47. Autologous dendritic cells (DC) are prepared from autologous PBMC exposed to sargramostim (GM-CSF), interleukin-4, and tumor necrosis factor alpha and pulsed with autologous tumor cell lysate. Patients receive autologous tumor cell lysate-pulsed DC IV over 5-10 minutes on days 0, 28, and 56.

Cohorts of 3-6 patients receive escalating doses of autologous tumor cell lysate-pulsed DC until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 33% of all patients experience dose-limiting toxicity.

Patients are followed at day 84 and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 3-20 patients will be accrued for this study within 3-20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed melanoma

  * Stage III (lymph node or in-transit metastases) or IV (systemic metastases) disease
* Patients with relapsed disease OR who failed prior immunotherapy or chemotherapy are eligible (but trial not restricted to relapsed or refractory disease)
* Tumor tissue available and properly stored for lysate preparation

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 75,000/mm^3

Hepatic

* AST ≤ 2 times upper limit of normal (ULN) (3 times ULN for liver metastases)
* Bilirubin ≤ 2 times ULN
* Hepatitis B surface antigen negative
* Hepatitis C negative

Renal

* Creatinine ≤ 2.0 times ULN

Immunologic

* No active infection
* No history of autoimmune disease, including any of the following:

  * Inflammatory bowel disease
  * Systemic lupus erythematosus
  * Scleroderma
  * Rheumatoid arthritis
  * Multiple sclerosis
* No allergy to aminoglycosides or streptomycin
* HIV negative

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No significant comorbid illness
* No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* At least 10 days since prior immunotherapy

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* At least 6 weeks since prior steroid therapy
* No concurrent corticosteroids

Radiotherapy

* At least 10 days since prior radiotherapy
* No concurrent radiotherapy

Surgery

* At least 10 days since prior surgery
* Prior diagnostic or palliative surgery allowed provided the patient has fully recovered

Other

* No concurrent immunosuppressive or potentially immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-02; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Ex Vivo Matured Dendritic Cell Therapy in Patients with Melanoma | 2005-2006

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P. Tretter, MD, Study Chair — Norris Cotton Cancer Center
Locations (1):
- Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States